CLINICAL TRIAL: NCT01547390
Title: Early Prediction and Aspirin for Prevention of Preeclampsia
Brief Title: Early Prevention of Preeclampsia Study
Acronym: EPAPP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated after Aspirin was recommended by the USPTF to Prevent Preeclampsia.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201112007
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Preeclampsia
Keywords: preeclampsia; Aspirin
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental): Aspirin 81mg one tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Interventions: Drug: Aspirin
- placebo (Placebo Comparator): placebo one tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aspirin
  Arms: Aspirin
Drug: placebo
  Arms: placebo

SUMMARY:
This is a randomized controlled trial to estimate the efficacy of low dose aspirin for preventing preeclampsia in women identified as high risk. The investigators hypothesize that the risk of preeclampsia in women identified by a first trimester multiparameter predictive model to be at high risk will be significantly reduced by initiating low dose aspirin early in pregnancy.

DETAILED DESCRIPTION:
This will be a randomized control trial to estimate the efficacy of low dose aspirin in preventing preeclampsia in women identified in the first trimester to be at high risk. We will also obtain maternal blood, cord blood and placenta specimen for basic science studies to attempt to dissect biological mechanisms of aspirin effects. In addition we will conduct a cost-benefit analysis to determine the cost effectiveness of screening and using aspirin prophylaxis for screen positive women.

Rationale for Design: The randomized control trial is the 'gold standard' of research design. Other designs such as case-control, retrospective cohort and prospective cohort are limited by potential bias and confounding. Randomly assigning subjects to different interventions minimizes selection bias. The random assignment also results in groups that are likely to be similar with regards to important confounding variables. This minimizes confounding by both measured and unmeasured factors. While random allocation does not guarantee the groups will be identical, it does ensure that any differences between them are due to chance alone. Finally, randomization produces groups that are random samples of the population. This permits use of standard statistical tests that are based on probability theory.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy undergoing ultrasound examination at 9 0/7 - 14 6/7 weeks
* any one or more factors identified as high risk from the identified risk factors: Chronic hypertension, prepregnancy diabetes mellitus, previous preeclampsia, obesity (BMI >30), bilateral uterine artery notches preeclampsia risk score greater than 6, low PAPP-A ( < 0.52 MoM)

Exclusion Criteria:

* Multiple gestations,
* fetal aneuploidy
* major fetal structural anomaly
* bleeding disorder
* allergy to aspirin
* women already on aspirin or heparin.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-03; Primary Completion 2015-07-20 (Actual); Study Completion 2015-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Odibo, MD, MSCE, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Odibo AO, Goetzinger KR, Odibo L, Tuuli MG. Early prediction and aspirin for prevention of pre-eclampsia (EPAPP) study: a randomized controlled trial. Ultrasound Obstet Gynecol. 2015 Oct;46(4):414-8. doi: 10.1002/uog.14889. Epub 2015 Aug 31. PMID 25914193

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1470 women screened, 138 were screen positive, and 53 consented to participate in the study and were randomized. Ten women in the aspirin group and 13 in the placebo group dropped out of the study.
Groups:
- Placebo: Study subjects receiving placebo one tablet orally per day
- Aspirin: Study subjects receiving aspirin 81 mg one tablet orally per day.
Period: Overall Study
Arm/Group | Placebo | Aspirin
Started | 27 | 26
Completed | 14 | 16
Not Completed | 13 | 10
Not completed — Withdrawal by Subject | 10 | 7
Not completed — termination of pregnancy | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 1 capsule orally daily
- Aspirin: 81mg, 1 capsule orally daily
- Total: Total of all reporting groups
Arm/Group | Placebo | Aspirin | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Maternal age at enrolment as reported by the participant
  years | 31.6 (6.1) | 30.0 (5.0) | 30.8 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 14 | 16 | 30
  Sex: Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 11 | 4 | 15
  White | 3 | 1 | 4
  Other | 0 | 11 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Preeclampsia
Description: Preeclampsia diagnosed per ACOG criteria: Blood pressure greater than 140/90 on 2 occasions 6 hrs apart and significant proteinuria (greater than 300mg in 24hrs).
Time Frame: within 3 months prior to delivery
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: 1 capsule orally, daily
Arm/Group | Placebo | Aspirin
Number analyzed (Participants) | 14 | 16
Participants | 3 | 3

2. Secondary Outcome: Number of Participants With IUGR, Early Preeclampsia, Severe Preeclampsia, Gestational Hypertension, Preterm Birth, Stillbirth, Placental Abruption, Antepartum Hemorrhage, Neonatal Death, NICU Admission, Miscarriage
Description: Intrauterine growth restriction (IUGR) - estimated fetal weight less than 10th percentile early preeclampsia - preeclampsia delivered prior to 34 weeks severe preeclampsia - blood pressure greater then 160/110 gestational hypertension - hypertension without features of preeclampsia preterm birth, stillbirth, placental abruption, antepartum hemorrhage, neonatal death, NICU admission, miscarriage.
  Statistical significance not reported due to the low recruitment and poor patient compliance.
Time Frame: within 3 months of delivery
Measure: Number; unit: participants
Arm/Group | Placebo | Aspirin
Number analyzed (Participants) | 14 | 16
participants
  Small for gestational age (IUGR) | 1 | 1
  Gestational hypertension | 0 | 2
  Early preeclampsia | 1 | 1
  Severe preeclampsia | 3 | 3
  Preterm birth | 2 | 1
  Stillbirth | 0 | 0
  Placental abruption | 0 | 0
  antepartum hemorrhage | 0 | 0
  neonatal death | 0 | 0
  NICU admission | 0 | 2
  miscarriage | 1 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Aspirin
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 3/14 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Aspirin (N=16)
Rash or hive (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated due to poor enrollment after Aspirin was recommended by the US Preventive Task Force for the Prevention of Preeclampsia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No